CLINICAL TRIAL: NCT02185352
Title: Randomized Phase II Study of Induction Bevacizumab, Etoposide and Cisplatin Followed by Whole Brain Radiotherapy (WBRT) Versus WBRT Alone in Breast Cancer With Untreated Brain Metastases
Brief Title: Bevacizumab, Etoposide and Cisplatin Followed by Whole Brain Radiotherapy in Breast Cancer With Brain Metastases
Acronym: A-Plus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201402059MIPD
Record Dates: First submitted 2014-06-25; First posted 2014-07-09 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Brain Metastases
Keywords: Bevacizumab; Brain Metastases; Breast Cancer; Chemotherapy; Whole Brain Radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Bevacizumab; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inductional BEEP regimen (Experimental): Induction BEEP regimen:
  Every 3 weeks a cycle for a total of 3 cycles (around 2 months)
  * Bevacizumab 15mg/kg IVF on D1
  * Etoposide 70 mg/m2 IVF QD, D2-4
  * Cisplatin 70 mg/m2 IVF on D2
  WBRT:
  3000cGy in 10 fractions
  Interventions: Drug: BEEP regimen
- WBRT alone (No Intervention): standard WBRT:
  3000cGy in 10 fractions

INTERVENTIONS:
Drug: BEEP regimen — Bevacizumab 15mg/kg IVF on D1, Etoposide 70 mg/m2 IVF QD, D2-4, Cisplatin 70 mg/m2 IVF on D2, repeat every 3 weeks, for 3 cycles
  Other Names: Bevacizumab; Etoposide; Cisplatin
  Arms: Inductional BEEP regimen

SUMMARY:
The primary objective of A-PLUS trial is to evaluate and compare the efficacy of induction BEEP (bevacizumab preconditioning followed by etoposide and cisplatin) followed by whole bran radiotherapy (WBRT) with WBRT alone in the controlling of brain metastases (BM) in metastatic breast cancer (MBC) patients who have not previously received WBRT.

In past 2 years, the research team has demonstrated that BEEP regimen is a highly effective treatment for brain metastases of breast cancer progressing from WBRT by a multi-center phase II study (ClinicalTrials.gov Identifier: NCT01281696). The basic concept of preconditioning, as referred to starting bevacizumab 1 day before chemotherapy, is that the effect of bevacizumab induced tumor vascular normalization takes time to mature.

The investigators hypothesized that as induction BEEP decreased the size of brain tumors, the effectiveness of WBRT would be maximized. The investigators expect this integrated approach will do greater benefit to MBC patients with BM, irrespective of subtype.

DETAILED DESCRIPTION:
Brain metastasis (BM) occurs in about 20% to 35% of metastatic breast cancer (MBC) patients. In contrast to recent advances in systemic treatment of MBC, there is much room for improvement in treatment of BM. At present, the standard treatment for inoperable/not suitable for radiosurgery BM is whole-brain radiotherapy (WBRT), but with only a median overall survival (OS) of 6 to 12 months and a high brain relapse rate ranging from 30% to 100%.

In MBC, 70% to 80% of patients with BM are presented with more than two brain metastatic tumors and are not candidate for both surgical treatment and stereotactic radiosurgery (SRS). Unlike patients with solitary or oligo-brain metastatic tumors, for whom the addition of local treatments such as surgery or SRS has been shown to improve OS and relapse rate; for patients with multiple brain metastases, WBRT remained the only standard treatment and improvements are desperately awaited.

Brain was once considered as a "sanctuary" area for systemic drugs due to the protection of blood-brain-barrier (BBB). Although some preclinical studies suggest that the BBB could be disrupted during the growth of brain metastatic tumor, the amount of chemotherapy drugs be delivered to brain tissue was still far lower than that could be achieved in serum. Bevacizumab, a vascular endothelial growth factor antibody, has shown the ability to "normalize" the peri-tumoral vessels in preclinical models. The investigators hypothesized that with the addition of bevacizumab, the chemotherapy drugs-etoposide and cisplatin, which were shown also to have some activity for BM-will be delivered more efficiently into the once "sanctuary" brain parenchyma, thus increasing the efficacy of BM treatment.

Recently, the research team have demonstrated that bevacizumab preconditioning followed by etoposide and cisplatin (BEEP) is a highly effective treatment for brain metastases of breast cancer progressing from radiotherapy by a multi-center phase II study. The basic concept of preconditioning, as referred to starting bevacizumab 1 day before chemotherapy, is that normalization effect takes time to mature. In that study, 35 patients were enrolled. Twenty seven patients (77.2%; 95%CI 59.9-89.6) achieved brain tumor volumetric response, defined as a ≥50% reduction in the volumetric sum of all measurable brain lesions in the absence of increasing steroid use, development of new brain lesion, or progressive neurologic symptoms. With a median follow-up of 11.0 months, the median CNS progression free survival (PFS) was 6.7 months (95% CI 5.1 to 8.3 months), and OS was 9.4 months (95% CI 7.3 to 11.5 months).

At present, lapatinib is the only molecular targeted agent proven effective for MBC patients with BM. The CNS response rate of first-line lapatinib plus capecitabine was 65% in WBRT-naïve, HER2-positive MBC patients with BM. However, the median CNS PFS is still disappointingly short at 5.5 months and the result is limited to MBC patients who are HER2-positive.

It has been demonstrated that brain tumor size is a predictor of WBRT failure. Given the high response rate of BEEP for BM in our phase II trial, the investigators hypothesized that as induction BEEP decreased the size of BM, the effectiveness of WBRT would also be enhanced. This integrated approach will do greater benefit to MBC patients with BM, irrespective of subtype. Hence, the investigators plan to conduct this randomized phase II trial to evaluate the efficacy of induction BEEP followed by WBRT.

Sub study of A-PLUS: A Integrated Study of MRI and PET of The Brain in Evaluation of Neurocognitive Outcomes of Patients with Brain Metastasis Treated by Radiotherapy and Chemotherapy.

The participants of A-PLUS trial may be enrolled in an additional study of this trial. This additional prospective study aims to investigate the neurocognitive outcomes of patients with brain metastases treated by radiotherapy and chemotherapy. The evaluations include neurocognitive assessments, serial MRI and FDG PET-CT (Integrated MR-PET) at before and after the study treatment. A total of 80 participants will be enrolled. The study protocol was approved by the NTUH REC, No. 201412046MINA.

ELIGIBILITY:
Inclusion criteria:

* A histological confirmed invasive breast cancer.
* At least one measurable brain metastatic tumor. If the measurable brain lesion has previously received stereotactic radiosurgery, the tumor must be a progressive lesion after radiosurgery.
* Patients who had not received WBRT.
* Patients with HER2/neu overexpression or amplification and had received trastuzumab before the diagnosis of BM will be allowed but will be informed about other available treatment options such as lapatinib plus capecitabine.
* Karnofsky performance score (KPS) higher or equal to 30%.
* Patients must have adequate organ function and marrow reserve measured within 14 days prior to randomization
* Age 20 to 75 years.
* Patient's life expectancy is more than 3 months.
* All women of childbearing potential must have a negative pregnancy test obtained within 72 hours before starting therapy.
* Patients with reproductive potential must use effective contraception (hormone or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after the completion of therapy.
* Patients (or a surrogate) must be able to comply with study procedures and sign informed consent.

Exclusion criteria:

* Prior therapy with bevacizumab, sorafenib, sunitinib, or other VEGF pathway-targeted therapy.
* Patients who have history of disease progression or disease developed during prior cisplatin treatment.
* Patients who had leptomeningeal metastasis, either diagnosed by brain imaging study or confirmed by cerebrospinal fluid cytology examination.
* Patients who are eligible for and willing to receive brain surgery or stereotactic radiosurgery (SRS) as the initial treatment of BM.
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* History of thrombotic disorders.
* Active gastrointestinal bleeding.
* Patients with a history of self-reported intra-cranial hemorrhage or evidence of bleeding in previous cranial imaging.
* Patients with clinical signs or symptoms of gastrointestinal obstruction and who require parenteral hydration and/or nutrition because of obstruction.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of first dose of bevacizumab.
* Clinically significant peripheral artery occlusive disease.
* Arterial thromboembolic event within the past 6 months, including transient ischemic attack, cerebrovascular accident, unstable angina, or myocardial infarction.
* History of gross hemoptysis (e.g., ≥ 1 teaspoon of bright red blood).
* Other malignancy within 5 years except cured basal cell or squamous cell skin cancer or carcinoma in situ of the cervix.
* Psychiatric illness or social situation that would preclude study compliance.
* Serious non-healing wound, ulcer, or bone fracture.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment.
* Prior minor surgery within 7 days.
* Concurrent chronic daily aspirin (> 325 mg/day), dipyridamole, ticlopidine, clopidogrel, cilostazol, non-steroidal anti-inflammatory agents known to inhibit platelet function.
* Concurrent therapeutic anticoagulation, but prophylactic anti-coagulation of venous access devices is allowed.
* History of allergic reaction to compounds of similar chemical composition to the study drugs.
* Pregnancy or lactation.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
The Brain-specific progression free survival (BS-PFS) | 2.5 years
  To evaluate and compare the brain-specific progression free survival (BS-PFS) of the two treatment arms based on RECIST 1.1.

SECONDARY OUTCOMES:
The 2-month brain-specific objective response rate (BS-ORR) | 2 months
  To compare the 2-month brain-specific objective response rate (BS-ORR) of the two treatment arms based on volumetric analysis (CNS composite response criteria).

OTHER OUTCOMES:
The BS-PFS based on volumetric analysis (CNS composite response criteria) | 2.5 years
  To compare the BS-PFS of the two treatment arms based on volumetric analysis (CNS composite response criteria).
The 8-month BS-PFSR based on volumetric analysis (CNS composite response criteria) | 8 months
  To compare the 8-month BS-PFSR of the two treatment arms based on volumetric analysis (CNS composite response criteria).
The BS-ORR based on volumetric analysis (CNS composite response criteria) | 5 months
  To evaluate and compare the BS-ORR of the two treatment arms based on volumetric analysis (CNS composite response criteria).
The 8-month BS-PFSR based on RECIST 1.1 | 8 months
  To compare the 8-month BS-PFSR of the two treatment arms based on RECIST 1.1.
The progression free survival (PFS) and overall survival (OS) | 2.5 years
  To observe the difference of the PFS and OS between the two treatment arms.
The extra-CNS tumor progression free survival (PFS) based on RECIST 1.1 | 2.5 years
  To evaluate and compare extra-CNS tumor progression free survival (PFS) of the two treatment arms (and followed by physician/investigator choice of systemic therapy) based on RECIST 1.1.
The time-to-improvement of neurological function | 3 months
  To evaluate the difference of time-to-improvement of neurological function between the two treatment arms.
Number of participants with adverse events | 3 months
  To evaluate and compare the safety profile of the two treatment arms according CTCAE 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, M.D, Ph.D., Principal Investigator — National Taiwan Unversity Hospital
Locations (8):
- Taiwan (8):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital-LinKou, Taoyuan District

REFERENCES:
- [Derived] Chen TW, Dai MS, Tseng LM, Chen SC, Chao TY, Chao TC, Chang YC, Chiu CF, Liu CT, Lin CH, Liu CY, Chen YF, Chang DY, Yu JC, Rau KM, Hsieh YY, Shen SC, Huang SM, Cheng AL, Lu YS. Whole-Brain Radiotherapy Alone vs Preceded by Bevacizumab, Etoposide, and Cisplatin for Untreated Brain Metastases From Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2024 Mar 1;10(3):325-334. doi: 10.1001/jamaoncol.2023.5456. PMID 38127335